CLINICAL TRIAL: NCT06524076
Title: Clinical and Radiographic Evaluation of Partial Pulpotomy Versus Complete Pulpotomy in Vital Pulp Therapy in Primary Molars Using NeoPUTTY™ (MTA): Randomized Clinical Trial
Brief Title: Evaluation of Success Rate of Partial Pulpotomy Versus Complete Pulpotomy in Primary Molars Using NeoPUTTY MTA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Yara Ayman, Internal resident of Pediatric Dentistry and Public Health, Cairo University, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 28052024
Record Dates: First submitted 2024-07-22; First posted 2024-07-29 (Actual); Last update posted 2024-08-14 (Actual); Status verified 2024-08

CONDITIONS: Pulp Disease, Dental
MeSH Terms: conditions — Dental Pulp Diseases

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Partial Pulpotomy (Experimental)
  Interventions: Procedure: Partial Pulpotomy
- Complete pulpotomy (Active Comparator)
  Interventions: Procedure: Complete pulpotomy

INTERVENTIONS:
Procedure: Partial Pulpotomy — After removing caries high-speed handpiece with water coolant using a round diamond bur. Once there is an exposure, the bur is changed with another sterile one with which the superficially inflamed pulp tissue will be gently removed to a depth of 1-3 mm beneath the pinpoint pulp exposure that occurred at the end of caries removal. A sterile cotton pellet with saline will be placed with light pressure for 2-3 minutes to achieve hemostasis.
  Arms: Partial Pulpotomy
Procedure: Complete pulpotomy — After removing caries with a large round bur, the access cavity will be opened. Excavation of inflamed coronal pulp tissues will be done using a sharp excavator. A sterile cotton pellet with saline will be placed with light pressure for 2-3 minutes to achieve hemostasis.
  Arms: Complete pulpotomy

SUMMARY:
Evaluating the clinical and radiographic success of partial pulpotomy compared to complete pulpotomy in vital primary second molars with reversible pulpitis using NeoPUTTY™ (MTA).

DETAILED DESCRIPTION:
Children with symptoms of reversible pulpitis in their second primary molar will be chosen to be enrolled in the study, and then randomly allocated into two groups. One group will undergo partial pulpotomy and the other group complete pulpotomy and followed up for 12 months. The blinding of the operator is not possible due to the nature of the technique used. Trial participants, outcome assessors and statistician will be blinded.

1. Informed consent from participating children's parents.
2. Baseline records photographs, percussion test, periapical radiograph and personal data collection.
3. Diagnostic chart with personal, medical and dental history will be filled.
4. Allocation (concealed by withdrawing a sealed opaque envelope containing Four-folded numbered papers containing the type of vital pulp therapy technique that will be used then writing the patient's name and I.D. on it and will be opened after removing the carious lesion).
5. Clinical examination will be performed to assess the clinical inclusion criteria. (Pulpal and periapical diagnoses are established after clinical examination).
6. Preoperative and Postoperative photographs will be taken.

ELIGIBILITY:
Inclusion Criteria:

* Patients:

  * Aged 4-7 years, in good general health and medically within normal.

Teeth:

* Restorable mandibular second primary molars.
* History of reversible pulpitis.

Preoperative radiograph:

* Absence of periapical or inter-radicular radiolucency.
* Absence of widening of periodontal ligaments (PDL) space.
* Absence of internal or external root resorption.

Exclusion Criteria:

* Patients:

  * With systemic disorders.
  * Physical or mental disabilities.
  * Unable to attend follow-up visits.
  * Refusal of Participation.
  * Refusal to sign the informed consent.

Teeth:

* Previously accessed teeth.
* Mobile mandibular second primary molar.
* Swelling in the vestibule or on palpation.
* Pain on percussion.

Ages: 4 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2024-09-22 (Estimated); Primary Completion 2024-12-22 (Estimated); Study Completion 2025-12-22 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain | one week postoperative
  Postoperative pain assessment through Visual Analog Scale (the lower the value the better).
Swelling/ Fistula | 3, 6, 9, 12 months
  Assessment of swelling and fistula through visual examination.
Mobility | 3, 6, 9, 12 months
  Assesment of pathological mobility using mobility test.

SECONDARY OUTCOMES:
Radiographic success | 0, 6, 12 months
  Radiographic evaluation (Radiolucency at furcation or periapical, internal or external root resorption) through visual interpretation of digital radiograph at 0, 6 and 12 months postoperatively.

CONTACTS AND LOCATIONS:
Overall Officials: Hany M. Saber, PHD, Study Chair — Faculty of Dental Medicine, Cairo University; Hanaa M. Abd El Moniem, PHD, Study Director — Faculty of Dental Medicine, Cairo University; Yara A. Badr, Masters, Principal Investigator — Faculty of Dental Medicine, Cairo University